CLINICAL TRIAL: NCT03480048
Title: Breastfeeding Support and Weight Management for Black Women: A Dual Intervention
Brief Title: Breastfeeding Support and Weight Management for Black Women
Acronym: MamaBear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jean Kerver, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC105989; 1R21HD085138-01A1 (NIH)
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Breastfeeding; Weight Loss
MeSH Terms: conditions — Breast Feeding; Weight Loss | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding and weight loss support (Experimental): Participants receive a combination of in-person, phone, and online support for breastfeeding and postpartum weight management.
  Interventions: Behavioral: Breastfeeding and weight loss support
- Usual care (No Intervention): Participants receive usual care from their prenatal care provider.

INTERVENTIONS:
Behavioral: Breastfeeding and weight loss support — The intervention is based on the Loving Support peer counseling breastfeeding model developed by the Special Supplemental Program for Women Infants and Children (WIC) with added components to promote postpartum weight loss.
  Arms: Breastfeeding and weight loss support

SUMMARY:
This study, in African American mothers in Detroit, will test an intervention that combines home visiting by experienced peer counselors with a smart phone-based weight control program. The investigators are trying to help mothers breastfeed their babies longer, and also help them get back to the weight they were before they were pregnant. This trial will help the investigators to guide policies in the state of Michigan and has the potential to improve the health of both mothers and babies everywhere.

DETAILED DESCRIPTION:
Excessive pregnancy-related weight retention is an important determinant of obesity and is more common among African American women. At the same time, breastfeeding, which has been recommended as a strategy to decrease weight retention is lowest among African American women. This racial disparity in breastfeeding may partly explain the disparity in obesity, but even if the two are not causally related, a dual intervention designed to increase breastfeeding duration and decrease postpartum weight retention makes practical sense because both are associated with the same critical postpartum time window.

For this study, the investigators will incorporate a postpartum weight management component into an effective breastfeeding support program. This dual intervention will use a combination of in-person, telephone, and interactive web/mobile-based health counseling to provide education and support for breastfeeding difficulties and postpartum weight management. The intervention will be delivered by peer counselors who will be trained to provide support using motivational interviewing techniques with consultation by experts. The investigators have designed the dual intervention to provide encouragement, information, and problem-solving assistance at the appropriate pre or postpartum stage for both breastfeeding support and maternal weight management. The mixed delivery mode has proven effective in other settings and is important to build a trusting relationship while allowing frequent and flexible methods for communicating during this vulnerable time in a new mom's life. The overall goal of this developmental/exploratory R21 proposal is to gather pilot data to effectively refine the intervention so that it can be tested in a larger, longer study using a factorial design in a future R01 phase. The investigators will recruit, in one large inner-city prenatal care clinic (Henry Ford Health System, Detroit, MI), pregnant African American women (32-36 weeks gestation) who are considering breastfeeding (n=80), randomize them to the intervention or to a usual care group, and follow all participants to 20 weeks postpartum. The specific aims are to: 1) test feasibility; 2) assess acceptability; and 3) estimate the effect size of the intervention at 20 weeks postpartum relative to the usual care group on (1) breastfeeding duration and (2) postpartum weight retention. This project is significant because the combined intervention is designed to work synergistically on two interrelated, highly prevalent problems that disproportionately disadvantage African American families.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, African American women, aged 18 and older, intending to breastfeed, ability to complete surveys in English

Exclusion Criteria:

* Contraindications to breastfeeding, high-risk pregnancy,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be pregnant.
Enrollment: 53 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Kerver, PhD, Principal Investigator — Michigan State University
Locations (1):
- Henry Ford Health System, New Center One Women's Clinic, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shipp GM, Weatherspoon LJ, Comstock SS, Norman GS, Alexander GL, Gardiner JC, Kerver JM. Breastfeeding Self-Efficacy as a Predictor of Breastfeeding Intensity Among African American Women in the Mama Bear Feasibility Trial. Breastfeed Med. 2022 May;17(5):453-458. doi: 10.1089/bfm.2021.0301. Epub 2022 Feb 15. PMID 35166571

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breastfeeding and Weight Loss Support | Usual Care
Started | 28 | 25
Completed | 18 | 17
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breastfeeding and Weight Loss Support | Usual Care | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 53
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 25 | 53
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Still Breastfeeding at 20 Weeks Postpartum
Description: Count of women who report any breastfeeding at 20 weeks postpartum
Time Frame: 20 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Breastfeeding and Weight Loss Support | Usual Care
Number analyzed (Participants) | 18 | 17
Participants | 9 | 8

2. Primary Outcome: Change in Weight From Baseline
Description: Weight at 20 weeks postpartum minus pre-pregnancy weight.
Time Frame: Baseline and 20 weeks postpartum
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Breastfeeding and Weight Loss Support | Usual Care
Number analyzed (Participants) | 18 | 17
pounds | 1.5 (19.2) | 11.7 (22.3)

ADVERSE EVENTS:
Time Frame: From study enrollment during late pregnancy through 20 weeks postpartum, or about 6-7 months.
Arm/Group | Breastfeeding and Weight Loss Support | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03480048/Prot_SAP_ICF_000.pdf